CLINICAL TRIAL: NCT02079779
Title: Study of the Effectiveness of an Interactive Robot for the Rehabilitation of the Upper Limb in Acute Stroke Patients by Evaluating the 3 Fields of the ICF: a Prospective, Randomized, Controlled, Simple Blind Study
Brief Title: Efficacy Study of an Interactive Robot for the Rehabilitation of the Upper Limb in Acute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IONS-Gilliaux-02
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Acute Stroke
Keywords: Robotic-assisted therapy; Acute Stroke; International Classification of Functioning, Disability and Health
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robotic-assisted therapy (Experimental): All patients will receive a similar classical rehabilitation as a basis. The 30 patients of this group will receive a supplement of robotic-assisted therapy.
  Interventions: Other: Robotic-assisted therapy; Other: Classical therapy
- Classical therapy (Active Comparator): All patients will receive a similar classical rehabilitation as a basis. The 30 patients of this group will receive a supplement of classical rehabilitation.
  Interventions: Other: Classical therapy

INTERVENTIONS:
Other: Robotic-assisted therapy — The robotic device is designed to intensively rehabilitate the upper limb. Indeed, this robot allows the patient to perform a lot of active, passive, or assisted exercises. The level of assistance is determined and provided by the robot in function of the patient performance (i.e. quality of movements).
  Arms: Robotic-assisted therapy
Other: Classical therapy — Conventional therapy will be performed by therapists specialized in neuro-rehabilitation

SUMMARY:
Stroke is the principal cause of permanent disability within the investigators population. This incapacity justifies an intensive and prolonged multidisciplinary rehabilitation, which can be optimized by robotics.

The investigators team has developed a robot designed to rehabilitate the upper limb. This robot allows the patient to perform active, passive, or assisted exercises. The system is also able to assess movement quality and to provide a feedback to the patient and the therapist via a graphical interface. This therapy is designed to improve functional recovery of patients, and then their quality of life.

Few quality studies have evaluated the efficacy of robotic assisted therapy in patients at the acute stage of rehabilitation (< 3 months post stroke) when most improvements are observed.

Thus, the aim of this study was to objectify the effectiveness of robotic-assisted rehabilitation in the acute stage after stroke by evaluating the 3 fields of the ICF (International Classification of Functioning, Disability and Health) and performing a prospective multicenter randomized controlled single blind trial. In this study, 60 stroke patients will be recruited and randomized into two groups. All patients will receive a similar classical rehabilitation as a basis. Patients of the control and experimental groups will receive a supplement of classical rehabilitation and robotic-assisted therapy, respectively.

DETAILED DESCRIPTION:
INTRODUCTION

The cerebral vascular accident affects two people per thousand each year (Duncan et al. 2005). This injury is the leading cause of permanent disability in our population. The brain damage is expressed by different neurological impairments and functional disabilities. These disabilities justify intensive and sustained multidisciplinary rehabilitation to reduce neurological impairments, to improve the activities and participation of patients, and, ultimately, their quality of life (Duncan et al., 2005).

Recently appeared in rehabilitation to stimulate maximum brain plasticity robotic devices meet the actual recommendations existing in stroke's rehabilitation (Langhorne et al., 2011). Indeed, the robots allow the execution of a large number of movements whose quality is controlled. A visual interface gives the patient a feedback of its movements, and offers exercises oriented functional tasks that have meaning for him and the possibly dive into a virtual reality. All these elements justify the clinical development of robots to assist the therapists (Pignolo et al. 2009).

The therapeutic efficacy of these robots for the rehabilitation of the upper limb was evaluated especially in chronic stroke patients (> 6 months after stroke) (Mehrholz et al., 2012). Unfortunately, few quality studies was conducted in these patients at the acute stage of rehabilitation, during which the potential of brain plasticity is the most important and the largest functional progress are observed (Stinear et al. 2012). In addition, few studies have evaluated the effect of these therapies robotic on the three fields of the ICF (Mehrholz et al., 2012). Many studies focus on impairments (e.g. muscle strength) without assessing the functional ability of the patient in activities of daily living.

OBJECTIVES

To perform a multicenter, single blind, randomized, controlled trial to assess the efficacy of of robotic-assisted therapy in acute stroke patients by evaluating the three fields of the ICF.

METHODS

Patients will be included in the Cliniques Universitaires Saint-Luc (Brussels, Belgique) and the center of William Lennox (Ottignies, Belgique). The patients will be randomised into two groups (control and experimental), using a stratified randomization method to ensure the equivalence of the two groups for motor neurological impairments (score of the Fugl-Meyer). This randomization will be organized independently in each centre participating in the study. The study of statistical power shows that 27 patients per group are necessary. This study of power has taken into account a statistical power desired to 99%, a minimum detectable change to 0.09 and a standard deviation of 0.08 on the upper limb kinematics of the patient (Gilliaux et al. 2014). In estimating a risk of out drop to 10%, the investigators plan to recruit 60 patients.

In each centre, in the acute phase, the patients receive daily a multidisciplinary rehabilitation (physiotherapy, occupational therapy, speech therapy,...) more or less intensive (60 to 300 min). In the experimental group, one of these daily therapies will be devoted to the rehabilitation robot, 4 times a week for 9 weeks. The control group will benefit from conventional treatments. As such, the duration of support will be similar between the two groups. All treatments will be administered by therapists specialized in neurological rehabilitation.

Patients will be evaluated three times in the study: before the start of treatments, at the end of treatments, and 6 months after the stroke event. All assessments will be carried out by a therapist which will be not informed the group that the patient is assigned (single-blind).

PERSPECTIVES

From this study, the investigators hope to demonstrate the efficacy of robotic-assisted therapy in acute stroke patients by evaluating the three fields of the ICF. These results could prove that this tool can be a significant complement for the stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* first stroke
* acute stroke (less than 1 month)
* unilateral localisation of the stroke
* moderate to severe upper limb impairments (7<Fugl Meyer score<50/66)

Exclusion Criteria:

* brainstem or cerebellum stroke
* an unstable clinical condition contraindicating the upper limb rehabilitation treatments
* cognitive disorders preventing the understanding of the instructions
* other neurological or orthopedic pathology affecting the upper limb

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01-09 (Actual); Primary Completion 2015-01-09 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Kinematic | Change from Baseline in Kinematic at an expected average of 2 months (after the treamtment) and 6 months post stroke

SECONDARY OUTCOMES:
Fugl-Meyer upper limb assessment | Change from Baseline in upper limb motor control at an expected average of 2 months (after the treamtment) and 6 months post stroke
Stroke Impairment Assessment Set (sensitive and Pain items) | Change from Baseline in sensitivity and pain at an expected average of 2 months (after the treamtment) and 6 months post stroke
Box and Block test | Change from Baseline in manual ability at an expected average of 2 months (after the treamtment) and 6 months post stroke
Strenght test of the Medical Research council | Change from Baseline in upper limb strenght at an expected average of 2 months (after the treamtment) and 6 months post stroke
Ashworth test | Change from Baseline in upper limb spasticity at an expected average of 2 months (after the treamtment) and 6 months post stroke
Bell's test | Change from Baseline in Hemineglect at an expected average of 2 months (after the treamtment) and 6 months post stroke
Wolf Motor Function Test | Change from Baseline in activity of daily living at an expected average of 2 months (after the treamtment) and 6 months post stroke
Abilhand | Change from Baseline in activity of daily living at an expected average of 2 months (after the treamtment) and 6 months post stroke
Activlim | Change from Baseline in activity of daily living at an expected average of 2 months (after the treamtment) and 6 months post stroke
Stroke Impact Scale (Participation item) | Change from Baseline in participation in social activities at an expected average of 2 months (after the treamtment) and 6 months post stroke

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Gilliaux, PhD student, Principal Investigator — Université Catholique de Louvain; Gaetan Stoquart, Professor, Principal Investigator — Université Catholique de Louvain; Christine Detrembleur, Professor, Principal Investigator — Université Catholique de Louvain
Locations (3):
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels
  - Centre Hospitalier Valida, Brussels
  - Centre Neurologique William Lennox, Ottignies

REFERENCES:
- [Background] Duncan PW, Zorowitz R, Bates B, Choi JY, Glasberg JJ, Graham GD, Katz RC, Lamberty K, Reker D. Management of Adult Stroke Rehabilitation Care: a clinical practice guideline. Stroke. 2005 Sep;36(9):e100-43. doi: 10.1161/01.STR.0000180861.54180.FF. No abstract available. PMID 16120836
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Mehrholz J, Hadrich A, Platz T, Kugler J, Pohl M. Electromechanical and robot-assisted arm training for improving generic activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD006876. doi: 10.1002/14651858.CD006876.pub3. PMID 22696362
- [Background] Pignolo L. Robotics in neuro-rehabilitation. J Rehabil Med. 2009 Nov;41(12):955-60. doi: 10.2340/16501977-0434. PMID 19841823
- [Background] Stinear CM, Barber PA, Petoe M, Anwar S, Byblow WD. The PREP algorithm predicts potential for upper limb recovery after stroke. Brain. 2012 Aug;135(Pt 8):2527-35. doi: 10.1093/brain/aws146. Epub 2012 Jun 10. PMID 22689909
- [Background] Gilliaux M, Lejeune TM, Detrembleur C, Sapin J, Dehez B, Selves C, Stoquart G. Using the robotic device REAplan as a valid, reliable, and sensitive tool to quantify upper limb impairments in stroke patients. J Rehabil Med. 2014 Feb;46(2):117-25. doi: 10.2340/16501977-1245. PMID 24213596